CLINICAL TRIAL: NCT01083784
Title: The Benefit of Prophylactic Anticonvulsant in Post Cardiac Arrest Syndrome With Induced Mild Hypothermia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: MS SIM, MD, Dept.of emergency medicine, Assistant professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-08-038
Record Dates: First submitted 2010-03-07; First posted 2010-03-10 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; Prophylactic anticonvulsant
MeSH Terms: conditions — Heart Arrest | interventions — Valproic Acid; Clonazepam; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylactic group (Experimental): the group that used prophylactic anticonvulsants (valproate, clonazepam)
  Interventions: Drug: Use of prophylactic anticonvulsants (valproate, clonazepam)
- Control group (No Intervention): control group
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Use of prophylactic anticonvulsants (valproate, clonazepam) — start at hypothermia induction valproate : 30mg/kg iv loading - 8hr after - 6mg/kg q 8hr iv till 72hr clonazepam : 1mg po bit via L-tube till 72 hr
  Arms: Prophylactic group
Drug: Control group — Control group
  Arms: Control group

SUMMARY:
Cardiac arrest is a leading cause of sudden death, but the survival rate of cardiac arrest is only 5-35%.

Although, the first resuscitation of cardiac arrest patient would be success, the hypoxic brain injury after cardiac arrest is an important cause of the mortality and the morbidity.

For the management of the hypoxic brain injury after cardiac arrest, American Heart Association and European Resuscitation Council recommend induced mild hypothermia therapy. And, ILCOR(International Liaison Committee on Resuscitation) announced the standard treatment of post cardiac arrest syndrome(the success state of first resuscitation of the cardiac arrest patient) included the induced mild hypothermia therapy at September, 2008.

The generalized seizure and myoclonus arise in over 60% of post cardiac arrest syndrome patients and they are very difficult to control. Also, the occurrence of them implies poor prognosis of the patient.

Although, mild hypothermia therapy could be decrease the development and propagation of generalized seizure and myoclonus theologically, the therapy could not prevent the development and propagation of them entirely. Therefore, the use of prophylactic anticonvulsant should be needed. But, there is not randomized control study about the use of prophylactic anticonvulsant.

We hypothesized that the use of prophylactic anticonvulsant to post cardiac arrest syndrome patients would decrease the rate of occurrence of generalized seizure and myoclonus and would improve the neurologic outcome.

We planed that we used two anti-epileptic drugs - valproate, clonazepam - for the prophylactic anticonvulsant. The valproate and clonazepam are in general use for prevention and treatment of generalized seizure and myoclonus and are recommended to treat of generalized seizure and myoclonus to post cardiac arrest syndrome patients by 2008 guideline of ILCOR.

ELIGIBILITY:
Inclusion Criteria:

* Age : over 18, under 80
* Witnessed arrest
* Successful first resuscitation (ROSC should be last for 20 min.)
* Coma or Semicoma state
* Mean arterial pressure > 60mmHg
* Peripheral Oxygen saturation > 85%
* Expected life span before cardiac arrest > 3 month.
* Performance scale before cardiac arrest > 3 month.

Exclusion Criteria:

* Cause of arrest

  * Sepsis, Progression of malignancy, Trauma, Hemorrhagic shock
* Known Coagulopathy
* Major operation within 7 days
* Previous seizure history
* current use of valproate or clonazepam

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
electroencephalogram (EEG) | 72hr after cardiac arrest
  Seizure activity will be measured by EEG EEG will be interpreted by Nerologist

SECONDARY OUTCOMES:
CPC score (cerebral performance category) score | 1month and 3 month after cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Min Seob Sim, Master, Principal Investigator — Dept. of Emergency Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] 1. Willis, C.D., et al., Cardiopulmonary resuscitation after traumatic cardiac arrest is not always futile. Injury, 2006. 37(5): p. 448-54. 2. Eisenberg, M.S., et al., Cardiac arrest and resuscitation: a tale of 29 cities. Ann Emerg Med, 1990. 19(2): p. 179-86. 3. Edgren, E., et al., Assessment of neurological prognosis in comatose survivors of cardiac arrest. BRCT I Study Group. Lancet, 1994. 343(8905): p. 1055-9. 4. Nolan, J.P., et al., Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication.Resuscitation, 2008. 79(3): p. 350-79. 5. Neumar, R.W., et al., Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication. Circulation, 2008. 118(23): p. 2452-83. 6. Kuboyama, K., et al., Delay in cooling negates the beneficial effect of mild resuscitative cerebral hypothermia after cardiac arrest in dogs: a prospective, randomized study. Crit Care Med, 1993. 21(9): p. 1348-58. 7. Weinrauch, V., et al., Beneficial effect of mild hypothermia and detrimental effect of deep hypothermia after cardiac arrest in dogs. Stroke, 1992. 23(10): p. 1454-62. 8. Sterz, F., et al., Mild hypothermic cardiopulmonary resuscitation improves outcome after prolonged cardiac arrest in dogs. Crit Care Med, 1991. 19(3): p. 379-89. 9. Leonov, Y., et al., Mild cerebral hypothermia during and after cardiac arrest improves neurologic outcome in dogs. J Cereb Blood Flow Metab, 1990. 10(1): p. 57-70. 10. Bernard, S.A., et al., Treatment of comatose survivors of out-of-hospital cardiac arrest with induced hypothermia. N Engl J Med, 2002. 346(8): p. 557-63.